CLINICAL TRIAL: NCT06853379
Title: Aromatherapy Versus Diet Management on Children with Primary Nocturnal Enuresis
Brief Title: Aromatherapy Versus Diet
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Cairo University (Other)
Responsible Party: Principal Investigator, Ahmed fekry ibrahim salman, assistant professor, Cairo University
Allocation: Randomized | Model: Crossover | Masking: Single | Purpose: Treatment
Other Study IDs: aromatherapy versus diet
Record Dates: First submitted 2025-02-27; First posted 2025-03-03 (Actual); Last update posted 2025-03-03 (Actual); Status verified 2025-02

CONDITIONS: Nocturnal Enuresis
MeSH Terms: conditions — Nocturnal Enuresis | interventions — Aromatherapy

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- group A (Experimental): Children were receive dietary recommendations or nonspecific dietary advices such as reducing fluid intake after 6 p.m. The list of dietary advices have been made reviewing literature and consisted in a list of recommended food, not recommended food at evening and not recommended food
  Interventions: Behavioral: dietary recommendations; Other: aroma therapy
- Group B (Experimental): GROUP B receive Harpal product
  Interventions: Behavioral: dietary recommendations; Other: aroma therapy

INTERVENTIONS:
Behavioral: dietary recommendations — . receive dietary recommendations or nonspecific dietary advices such as reducing fluid intake after 6 p.m. The list of dietary advices have been made reviewing literature and consisted in a list of recommended food, not recommended food at evening and not recommended food
Other: aroma therapy — the case receive aroma therapy

SUMMARY:
Eligible children were randomly divided into 2 groups assigned to receive dietary recommendations (group A) or to receive herbal compounds (group B). Children were treated for a period of one week , then cross over the two groups is done

ELIGIBILITY:
Inclusion Criteria:

* The participants age will be ranged from 5to 10 years.
* primary Nocturnal enuresis(NE) number of wet nights/week is more than 4\7

Exclusion Criteria:

* secondary nocturnal enuresis to any neurological disorders , musculoskeletal problems, or congenital abnormalities
* the child receives any Pharmacological treatment to NE

Ages: 5 Years to 10 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 30 (Estimated)
Dates: Start 2025-03-05 (Estimated); Primary Completion 2025-05-05 (Estimated); Study Completion 2025-05-10 (Estimated)

PRIMARY OUTCOMES:
number of wet days per week | ; for baseline evaluation of number of wet days per week, if the number is less than 4\7 the child will be excluded from the study. Second week; group A receives dietary recommendations , group B receives herbal compounds
  for baseline evaluation of number of wet days per week, if the number is less than 4\7 the child will be excluded from the study.

IPD SHARING:
Plan to Share IPD: Undecided